CLINICAL TRIAL: NCT06726343
Title: Maternal Fetal Device Performance Testing During Antepartum Singleton Monitoring
Brief Title: Maternal Fetal Device Performance Singleton
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SA-000072
Record Dates: First submitted 2024-10-28; First posted 2024-12-10 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Singleton

STUDY DESIGN:
Intervention Model Description: Pregnant women of ≥22 weeks gestation will undergo two 30-minute monitoring sessions (60 minutes total). One with currently approved Corometrics 259cx and one with the investigational device. During both monitoring sessions, maternal pulse rate will be monitored using SpO2 and the investigator shall be present to adjust the transducer placement as needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: 22 0/7 - 24 6/7 Weeks (Active Comparator): All subjects will undergo the same interventions as part of the study procedures but will be divided into groups based on gestational age groups. Each study subject will undergo two 30-minute monitoring sessions (60 minutes total). One with FDA approved device and one with the investigational device. During both monitoring sessions, maternal pulse rate (MPR) will be monitored using SpO2 and the investigator shall be present to adjust the transducer placement as needed
  Interventions: Device: Fetal Monitoring Device; Device: Investigational Fetal Monitoring Device
- Group 2: 25 0/7 - 31 6/7 Weeks (Active Comparator): All subjects will undergo the same interventions as part of the study procedures but will be divided into groups based on gestational age groups. Each study subject will undergo two 30-minute monitoring sessions (60 minutes total). One with FDA approved device and one with the investigational device. During both monitoring sessions, maternal pulse rate (MPR) will be monitored using SpO2 and the investigator shall be present to adjust the transducer placement as needed.
  Interventions: Device: Fetal Monitoring Device; Device: Investigational Fetal Monitoring Device
- Group 3: Greater than or equal to 32 0/7 Weeks (Active Comparator): All subjects will undergo the same interventions as part of the study procedures but will be divided into groups based on gestational age groups. Each study subject will undergo two 30-minute monitoring sessions (60 minutes total). One with FDA approved device and one with the investigational device. During both monitoring sessions, maternal pulse rate (MPR) will be monitored using SpO2 and the investigator shall be present to adjust the transducer placement as needed.
  Interventions: Device: Fetal Monitoring Device; Device: Investigational Fetal Monitoring Device

INTERVENTIONS:
Device: Fetal Monitoring Device — Fetal monitoring device is a multi-parameter maternal fetal monitor that is intended to monitor, store, display, transmit, and generate alarms for non-invasive and invasive clinical parameters of pregnant women and fetuses (singleton and twin), during the antepartum, intrapartum, and postpartum period.
  Other Names: Corometrics 259cx
Device: Investigational Fetal Monitoring Device — Fetal monitoring device is a multi-parameter maternal fetal monitor that is intended to monitor, store, display, transmit, and generate alarms for non-invasive and invasive clinical parameters of pregnant women and fetuses (singleton and twin), during the antepartum, intrapartum, and postpartum period.

SUMMARY:
Maternal Fetal Monitoring devices assist the health care professional in acquiring, monitoring, and storing fetal and maternal physiologic data which supports the decision making for pregnant women and the overall fetal health status during pregnancy and delivery. This study aims to support a new maternal fetal monitoring device with clinical data to demonstrate the equivalent performance against the currently marketed Corometrics 259cx. The fetal heart rate and will be collected during antenatal monitoring using standard of care Doppler ultrasound.

DETAILED DESCRIPTION:
This study aims to compare a maternal fetal monitoring device to the currently marketed Corometrics 259cx. Fetal heart rate and Fetal Movement Detection data will be collected during antenatal monitoring using standard of care Doppler Ultrasound transducers.

The new Maternal/Fetal Monitor is capable of monitoring heart rates (maternal/ fetal), maternal uterine contractions, as well as maternal blood pressure and maternal pulse oximetry. This study will compare clinical data between the current and the new monitor on non-laboring singleton gestation women.

Funding for this study will be provided by GE HealthCare. This study does not include patient advisors.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Singleton pregnancy.
3. Aged 18+.
4. Greater than or equal to 22 0/7 weeks gestation.
5. Patient has none of the exclusion criteria.

Exclusion Criteria:

1. Multiple pregnancy.
2. Involvement in another clinical trial currently or previously in this pregnancy that, in the investigator's opinion, would affect the conduct of this study.
3. Medical or obstetric problem that in investigator's opinion would make the patient incapable of taking part in the study.
4. Inability to understand the consent information due to medical illness, diminished intellectual capacity, or insurmountable language barrier.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Rabanal, NP, Principal Investigator — Element Materials Technology
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Euliano TY, Darmanjian S, Nguyen MT, Busowski JD, Euliano N, Gregg AR. Monitoring Fetal Heart Rate during Labor: A Comparison of Three Methods. J Pregnancy. 2017;2017:8529816. doi: 10.1155/2017/8529816. Epub 2017 Mar 14. PMID 28392944

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.08) | 30.3 (3.8) | 31.7 (3.65) | 31.07 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 9 | 8 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 10 | 9 | 10 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Height [Mean (Standard Deviation); unit: centimeters] | 64.6 (1.96) | 65.3 (3.23) | 64.5 (2.68) | 64.8 (2.61)
Weight [Mean (Standard Deviation); unit: pounds] | 157.8 (18.96) | 180.3 (55.02) | 176.2 (25.04) | 171.43 (36.67)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.69 (3.88) | 29.94 (9.71) | 29.86 (4.64) | 28.83 (6.56)

OUTCOME MEASURES:

1. Primary Outcome: Success Rate Calculated Based on Collection of Fetal Heart Rate Data From Investigational Devices on Subjects Enrolled in Each Gestational Age Group
Description: Collection of the presence of fetal heart rate rhythm data from the investigational device on subjects enrolled in each gestational age group to evaluate non-Inferiority in terms success rate which was defined as percentage of time in which the device gave FHR reading during the study monitoring period.
Time Frame: 30 minutes with investigational device over the course of 1 visit.
Population: The test was performed using two-sided 95% CI of the difference in Mean Success Rate (SR) for each gestational age group. Success rate is defined as percentage of time in which the device gave FHR reading during the study monitoring period.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- Group 1: 22 0/7 - 24 6/7 Weeks: Subjects with gestational ages between 22 weeks and 0/7 days and 24 weeks and 6/7 days.
- Group 2: 25 0/7 - 31 6/7 Weeks: Subjects with gestational ages between 25 weeks and 0/7 days and 31 weeks and 6/7 days.
- Group 3: Greater Than or Equal to 32 0/7 Weeks: Subjects with gestational age greater than 32 weeks and 0/7 days.
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
percentage | 85.01 [77.51 to 92.50] | 92.27 [86.51 to 98.03] | 98.43 [97.3 to 99.57]

2. Primary Outcome: Success Rate Calculated Based on Collection of Fetal Heart Rate Data From Coro 259cx Devices on Subjects Enrolled in Each Gestational Age Group
Description: Collection of the presence of fetal heart rate rhythm data from the Coro 259cx device on subjects enrolled in each gestational age group to evaluate non-Inferiority in terms success rate which was defined as percentage of time in which the device gave FHR reading during the study monitoring period.
Time Frame: 30 minutes with Coro 259cx over the course of 1 visit.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
percentage | 83.77 [74.41 to 93.13] | 89.07 [77.06 to 100] | 92.62 [88.27 to 96.96]

3. Primary Outcome: Difference in Success Rate Calculated Based on Collection of Fetal Heart Rate Data From Investigational and Coro 259cx Devices on Subjects Enrolled in Each Gestational Age Group
Description: Collection of the difference in the presence of fetal heart rate rhythm data sets from the Investigational and Coro 259cx devices on subjects enrolled in each gestational age group to evaluate non-Inferiority in terms success rate which was defined as percentage of time in which the device gave fetal heart rate reading during the study monitoring period. Difference in success rate was calculated as investigation minus Coro 259cx.
Time Frame: 30 minutes with Coro 259cx and 30 minutes of investigational over the course of 1 visit.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
percentage | 1.23 [-7.74 to 10.20] | 3.20 [-4.66 to 11.06] | 5.82 [2.14 to 9.50]

4. Secondary Outcome: Number of Raw Datasets of the Presence of Fetal Heart Rate During Continuous Monitoring Data From Investigational Device
Description: Collection of the number of raw data sets of fetal heart rate data sets for each group for internal testing purposes. No additional analysis was performed outside the success rate described in primary outcome.
Time Frame: 30 minutes with investigational device over the course of 1 visit.
Population: No subgroup analysis was performed.
Measure: Number; unit: data sets
Groups:
- Group 1: 22 0/7 - 24 6/7 Weeks: Subjects with gestational age between 22 weeks and 0/7 days and 24 weeks and 6/7 days.
- Group 2: 25 0/7 - 31 6/7 Weeks: Subjects with gestational age between 25 weeks and 0/7 days and 31 weeks and 6/7 days.
- Group 3: Greater Than or Equal to 32 0/7 Weeks: Subjects with gestational age greater than or equal to 32 weeks and 0/7 days.
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
data sets | 10 | 10 | 10

5. Secondary Outcome: Number of Raw Datasets of Automated Fetal Movement Detection and Remote Event Marks Data Sets on Investigational Device
Description: The collection of the number of raw data sets of automated fetal movement detection and remote event marks data sets per subject during continuous fetal monitoring from the investigational device on enrolled subjects for device validation. No analysis was performed on this data and it was collected for future testing purposes.
Time Frame: 30 minutes with investigational device over the course of 1 visit.
Population: No subgroup analysis was performed.
Measure: Number; unit: data sets
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
data sets | 10 | 10 | 10

6. Secondary Outcome: Number of Adverse Safety Events With Investigational Device
Description: The collection of the number of adverse events, serious adverse events, and/or device deficiencies reported on all enrolled subjects in the study using the investigational device.
Time Frame: 30 minutes with investigational device over the course of 1 visit.
Population: No AEs occurred during this study with the investigational device.
Measure: Number; unit: safety events
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
safety events | 0 | 0 | 0

7. Secondary Outcome: Number of Adverse Safety Events With Coro259 cx, FDA Approved Device
Description: The collection of the number of adverse events, serious adverse events, and/or device deficiencies reported on all enrolled subjects in the study using the FDA approved device.
Time Frame: 30 minutes with FDA approved device over the course of 1 visit.
Population: No AEs occurred during this study with the FDA approved device.
Measure: Number; unit: safety events
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
safety events | 0 | 0 | 0

8. Secondary Outcome: The Number of Raw Datasets of Automated Fetal Movement Detection and Remote Event Marks Data Sets on Coro 259cx Device
Description: as for outcome 5
Time Frame: 30 minutes with Coro 259cx, FDA approved device over the course of 1 visit.
Population: No subgroup analysis was performed.
Measure: Number; unit: data sets
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
Number analyzed (Participants) | 10 | 10 | 10
data sets | 10 | 10 | 10

ADVERSE EVENTS:
Time Frame: Duration of monitoring; approximately 60 minutes
Description: All adverse events (AE), including all serious adverse events (SAE), are required to be collected, investigated, and documented. AEs will be collected from [describe the reporting period, e.g., from the time they enter the scan room to the time they leave the scan room]. All AEs will be followed through to their resolution.
Arm/Group | Group 1: 22 0/7 - 24 6/7 Weeks | Group 2: 25 0/7 - 31 6/7 Weeks | Group 3: Greater Than or Equal to 32 0/7 Weeks
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT06726343/Prot_SAP_000.pdf